CLINICAL TRIAL: NCT06480409
Title: Program for Improving Students' Mental Health Using Virtual Reality - a Solution or a White Elephant?
Brief Title: **Virtual Reality in Student Mental Health: Solution or White Elephant?**
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Opole University of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Opole
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Mental Health Issue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR-based intervention (Experimental): The intervention group will participate in a structured VR-based relaxation program designed to improve mental health and reduce stress levels. The sessions will take place in a dedicated relaxation room equipped with immersive VR headsets and physiological sensors.
  Intervention Procedure:
  Duration and Frequency: Participants will engage in 15-minute VR relaxation sessions, held five times a week over a period of one month.
  VR Content: The VR sessions will feature high-quality 360° videos with therapeutic audio, including guided relaxation, calming music, and nature sounds.
  Interventions: Other: VR Mindfulness and Stress Reduction Program

INTERVENTIONS:
Other: VR Mindfulness and Stress Reduction Program — Intervention Procedure:
  Duration and Frequency: Participants will engage in 15-minute VR relaxation sessions, held five times a week over a period of one month.
  VR Content: The VR sessions will feature high-quality 360° videos with therapeutic audio, including guided relaxation, calming music, and nature sounds.
  Physiological Monitoring: Throughout the sessions, participants' physiological responses will be monitored using Polar H-10 sensors to measure heart rate variability (HRV), providing data on autonomic nervous system activity.
  Psychological Assessment: Participants will complete the Perceived Stress Scale (PSS-10) before and after the intervention to evaluate changes in stress levels.
  Cybersickness Monitoring: The occurrence of any adverse effects, such as cybersickness, will be monitored and recorded.

SUMMARY:
The COVID-19 pandemic drastically altered social structures, leading to prolonged isolation and remote learning for students, causing significant mental health issues. This project at Opole University of Technology aims to address these challenges through a virtual reality (VR)-based therapeutic program.

Objectives:

The project will utilize immersive VR technology to conduct relaxation sessions, creating a dedicated relaxation room equipped with VR headsets and physiological sensors. The goal is to assess the impact of VR-based therapy on students' autonomic nervous system and psychological well-being.

Key Hypotheses:

VR relaxation sessions will induce physiological relaxation. A 15-minute VR session will not cause cybersickness. Weekly VR sessions will reduce stress levels among students.

Methodology:

Using Polar H-10 sensors, the project will measure heart rate variability (HRV) to evaluate autonomic responses. Psychological stress will be monitored using the Perceived Stress Scale (PSS-10). A sample size of 50 participants, calculated with G*Power software, will be studied using repeated measures ANOVA.

DETAILED DESCRIPTION:
Project Objective and Scope:

The COVID-19 pandemic, declared by the World Health Organization in March 2020, significantly altered social structures globally. In Poland, the pandemic led to prolonged periods of physical isolation and remote learning for students, disrupting conventional educational routines and causing elevated levels of loneliness and mental health issues, particularly depression. Research indicates that 30% of students exhibited symptoms of depression, and 50% experienced heightened stress during the pandemic. This project aims to address these mental health challenges by implementing a virtual reality (VR)-based therapeutic program for students at Opole University of Technology.

Project Description:

The proposed project focuses on using immersive VR technology to conduct relaxation sessions for students. The initiative will create a relaxation room equipped with VR headsets and physiological sensors to monitor students' responses during VR sessions. The primary goal is to evaluate the impact of VR-based relaxation therapy on the autonomic nervous system and psychological well-being of students.

Specific Objectives:

Implementing VR in Medical Practice:

VR technology has proven effective in various medical fields, including surgery, rehabilitation, and mental health. This project will leverage immersive VR to create an engaging and effective therapeutic environment. The therapy sessions will be conducted using portable VR headsets, providing students with an immersive experience that isolates them from real-world stressors.

Scientific Analysis:

Physiological data will be collected using Polar H-10 sensors to assess heart rate variability (HRV), a measure of autonomic nervous system activity. This data will help determine the effectiveness of different VR scenarios in inducing relaxation and improving mental well-being. The project will also monitor psychological changes using the Perceived Stress Scale (PSS-10).

Methodology:

A sample size of 50 participants has been calculated based on previous studies using G*Power software. The study will use repeated measures ANOVA to analyze the data, ensuring robust statistical analysis. The project also plans to promote participation through local media, aiming to include students from various higher education institutions in the Opole region.

ELIGIBILITY:
Inclusion Criteria:

* acceptance to participate in the research
* age 19-30

Exclusion Criteria:

* diagnosed neurological diseases,
* fear of wearing goggles
* diagnosed diseases or injuries of the musculoskeletal system

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Physiological Relaxation | 20 min
  Participants will be monitored via heart rate variability (HRV) indicating a balanced autonomic nervous system response.
Stress Levels | 10 min
  Participants will be examined by the Perceived Stress Scale (PSS-10).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Education and Physiotherapy, Opole University of Technology, Opole, Poland

IPD SHARING:
Plan to Share IPD: No